CLINICAL TRIAL: NCT00308204
Title: Discoid Lupus Erythematosus of the Scalp and a Trial of Biologic Therapy With Raptiva
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: inadequate number of enrolled study subjects
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilma F. Bergfeld, Staff, The Cleveland Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACD3433s
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Discoid Lupus Erthematosus of the Scalp
Keywords: discoid lupus; lupus; discoid lupus erythematosus; lupus of the scalp
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — efalizumab

ARMS (1):
- Raptiva (Experimental): raptiva injection
  Interventions: Drug: Raptiva

INTERVENTIONS:
Drug: Raptiva — injection
  Other Names: efalizumab

SUMMARY:
The purpose of this study is to investigate the efficacy of Raptiva (efalizumab) in the treatment of discoid lupus erythematosus (DLE). Discoid lupus erythematosus is a chronic disorder, which may lead to permanent and progressive loss of hair. Lupus is a condition of chronic inflammation cause by an autoimmune disease. Autoimmune diseases are illnesses which occur when the body's tissues are attacked by its own immune system. The immune system is a complex system within the body that is designed to fight infectious agents, for example, bacteria, and other foreign invaders.

One of the mechanisms that the immune system uses to fight infections is the production of antibodies. Patients with lupus produce abnormal antibodies in their blood that target tissues within their own body rather than foreign infectious agents. Lupus can cause disease of the skin, heart, lungs, kidneys, joints, and nervous system. When only the skin is involved, the condition is called discoid lupus erythematosus (DLE).

Raptiva (efalizumab) is a humanized immunoglobulin(a protein extract from blood which fights off infection-sometimes called "antibody"), which targets the immune cells that are activated in inflammation. Raptiva has been approved for use in the management of psoriasis at doses of 1mg/kg, but is not approved for the treatment of DLE.

DETAILED DESCRIPTION:
This is an open label study in which the subject will be given the medication Raptiva (efalizumab) and they will be taught to self-inject by the dermatology nurse or research doctor. The subject will be administering 0.7mg/kg at week one and 1mg/kg once a week thereafter until week 24. If the subject feels uncomfortable self-administering these injections, the subject may identify a caregiver to administer these injections for them. He or she will be taught to administer these injections by the dermatology nurse or research doctor.

ELIGIBILITY:
Inclusion Criteria:

* adults with discoid lupus erythematosus with active area of disease involving at least 10% of scalp, confirmed by biopsy, bacterial and fungal culture negative.
* ability to provide written informed consent and comply with study assessments for the full duration of the study.
* adults 18 to 70 years of age.
* if a female of childbearing potential, a negative pregnancy test and commitment to the use of two forms of effective contraception (birth control) for the duration of the study are necessary.
* if a non-sterile male, commitment to the use of two forms of effective contraception (birth control) for the duration of the study is necessary.
* Platelets >100,000

Exclusion Criteria:

* subjects with known hypersensitivity to Raptiva (efalizumab) or any of its components
* pregnant or lactating women
* patients receiving immunosuppressive agents (not allowed 30 days or 5 half-live periods before Day 0, whichever is longer).
* prior enrollment in the study
* any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* participation in another simultaneous medical investigation or trial
* history of malignancy in the last 10 years.
* signs or symptoms of systemic lupus erythematosus.
* have a history of active tuberculosis or are currently undergoing treatment for tuberculosis. A purified protein derivative (PPD) test or chest x-ray will be performed at the screening visit. Patients with a positive PPD test or chest x-ray will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Efficacy in growing scalp hair | 36 weeks
  A 10% increase in visualized hair count in the target region between baseline and week 24 as determined by macrophotography and validated computer assisted dot mapping technique.

SECONDARY OUTCOMES:
clinical improvement of disease | 36 weeks
  Physician's global assessment (PGA) will be used to assess improvement of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Wilma F Bergfeld, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No